CLINICAL TRIAL: NCT01122784
Title: A Phase 2b Randomized, Single-Blinded Study to Evaluate the Safety and Immunogenicity of 80 µg Recombinant Plague Vaccine (rF1V) With and Without Adjuvant at Two Vaccination Schedules in Healthy Adult Volunteers
Brief Title: Randomized Single-Blinded Study to Evaluate Safety and Immunogenicity of Recombinant Plague Vaccine With and Without Adjuvant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: DynPort Vaccine Company LLC, A GDIT Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: rF1V-02b
Record Dates: First submitted 2010-05-07; First posted 2010-05-13 (Estimated); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Plague Vaccine
Keywords: Plague; Vaccine
MeSH Terms: conditions — Plague | interventions — Adjuvants, Pharmaceutic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 (Active Comparator): 160 Volunteers will be vaccinated with 80 mcg rF1V vaccine with adjuvant at Study Days 0, 56 and 182
  Interventions: Biological: rF1V vaccine (with Adjuvant)
- Group 2 (Active Comparator): 40 Volunteers will be vaccinated with 80 mcg rF1V vaccine without adjuvant at Study Days 0, 56 and 182
  Interventions: Biological: rF1V vaccine (without Adjuvant)
- Group 3 (Active Comparator): 160 Volunteers will be vaccinated with 80 mcg rF1V vaccine with adjuvant at Study Days 0, 56 and 121
  Interventions: Biological: rF1V vaccine (with Adjuvant)
- Group 4 (Active Comparator): 40 Volunteers will be vaccinated with 80 mcg rF1V vaccine without adjuvant at Study Days 0, 56 and 121
  Interventions: Biological: rF1V vaccine (without Adjuvant)

INTERVENTIONS:
Biological: rF1V vaccine (with Adjuvant) — 80 mcg rF1V vaccine with adjuvant given by intramuscular (IM) injection into the arm on Study Days 0, 56 and 182
  Other Names: Recombinant Plague Vaccine rF1V
  Arms: Group 1
Biological: rF1V vaccine (without Adjuvant) — 80 mcg rF1V vaccine without adjuvant given by intramuscular (IM) injection into the arm on Study Days 0, 56 and 182
  Other Names: Recombinant Plague Vaccine rF1V without Adjuvant
  Arms: Group 2
Biological: rF1V vaccine (with Adjuvant) — 80 mcg rF1V vaccine with adjuvant given by intramuscular (IM) injection into the arm on Study Days 0, 56 and 121
  Other Names: Recombinant Plague Vaccine rF1V
  Arms: Group 3
Biological: rF1V vaccine (without Adjuvant) — 80 mcg rF1V vaccine without adjuvant given by intramuscular (IM) injection into the arm on Study Days 0, 56 and 121
  Other Names: Recombinant Plague Vaccine rF1V without Adjuvant
  Arms: Group 4

SUMMARY:
Multicenter, randomized, single-blinded comparison of two formulations of the rF1V vaccine at a single dosage of 80 µg and two 3-dose schedules in 400 healthy, adult volunteers in four parallel cohorts. Two rF1V vaccine cohorts (N=160 each) and two rF1V antigen-only cohorts (N=40 each) will be vaccinated at two different three-dose schedules (Days 0, 56 and 182 or Days 0, 56 and 121).

DETAILED DESCRIPTION:
The objectives of this trial are: to compare the safety of rF1V vaccine administered in two different schedules through 28 days after each vaccination and cumulatively to Day 210; to compare the immunogenicity of rF1V vaccine administered in two different schedules through 28 days after Vaccination 3; to compare the safety and immunogenicity of rF1V vaccine administered by two different schedules through 12 months after Vaccination 3; and to assess the contribution of the adjuvant to the immunogenicity of the rF1V antigen.

ELIGIBILITY:
Inclusion Criteria:

1. The volunteer has signed the ICF and the HIPAA authorization and has successfully completed (at least 90% correct) the Test of Understanding.
2. The volunteer is a male or female 18 to 55 years of age (inclusive) at the time of the screening visit.
3. The volunteer is in good health as determined by the screening physician based upon medical history and physical examination, including vital signs within acceptable ranges.
4. The volunteer has acceptable ranges for the laboratory parameters.
5. The volunteer has no clinically significant abnormalities on ECG.
6. The volunteer agrees not to donate blood, plasma or blood components for therapeutic or research purposes, except to meet requirements of this study, at any time during the course of the study.
7. The volunteer is willing to have his or her blood samples stored for future plague research studies.
8. The volunteer is willing to comply with the requirements of the protocol through the end of the study.
9. Female volunteers must be of non-childbearing potential or, if of childbearing potential, must not be pregnant or lactating and must use acceptable contraception.

Exclusion Criteria:

1. History of plague exposure or disease or previous vaccination with any plague vaccine.
2. History of allergy to kanamycin or other aminoglycosides (e.g., gentamicin, tobramycin, amikacin).
3. History of anaphylaxis or other serious adverse reactions to vaccines or aluminum.
4. Active tuberculosis or other systemic infectious process by review of systems and PE.
5. History of chronic illness requiring continuous or frequent medical intervention or acute/chronic untreated conditions, multiple sclerosis, immunodeficiency, autoimmune or immunosuppressive disease or use of immunosuppressive medications.
6. Diabetes mellitus of any type requiring treatment with insulin or oral hypoglycemic drugs.
7. History of chronic, severe or recurrent joint pain (four or more clinically significant occurrences per year requiring treatment for remission) or arthritis of any etiology other than osteoarthritis.
8. Previous diagnosis of any serious psychiatric disorder.
9. Acute illness, evidence of significant active infection or evidence of systemic disease at the time of enrollment.
10. Oral temperature > 99.5°F.
11. Receipt of chemotherapeutic and immunosuppressive agents, including high-dose systemic glucocorticoids (i.e., prednisone-equivalent dose of > 20 mg/day).
12. Receipt of blood, any blood product or immune globulin.
13. Receipt of any investigational drug therapy or investigational implantable device or intent to receive any other investigational drug therapy or device throughout their study participation.
14. Receipt of any investigational vaccine.
15. Receipt or intent of any licensed nonliving vaccine.
16. Receipt of any licensed live vaccine within 60 days before Vaccination 1
17. Donation of more than 400 mL of blood 8 weeks before Vaccination 1.
18. Occupational or other responsibilities that would prevent completion of participation in the study.
19. Weight or body mass index (BMI) outside acceptable ranges.
20. Positive screening laboratory test for HIV antibody, HCV antibody or HBsAg.
21. A positive result on a urine drug screen that tests for common substances of abuse.
22. Female volunteer is pregnant or lactating.
23. The volunteer is currently on active duty in the U.S. military, or a member or relative of the clinical site study staff.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 402 (Actual)
Dates: Start 2010-07; Primary Completion 2012-05 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
To measure frequency and severity of local and systemic adverse events (AEs) through 28 days after each vaccination and cumulatively through Day 210. | Day 210 for Cohorts 1 through 4

SECONDARY OUTCOMES:
To assess the frequency and severity of local and systemic AEs of rF1V vaccine with and without adjuvant administered at 2 dosing schedules. | Through Day 540 for Cohort 1 and 2 and Day 485 for Cohorts 3 and 4.
To measure the proportion of volunteers in each cohort demonstrating seroconversion to vaccine antigens and the magnitude of the immune response. | Through Day 540 for Cohort 1 and 2 and Day 485 for Cohorts 3 and 4.

CONTACTS AND LOCATIONS:
Overall Officials: George Saviolakis, MD, Study Director — DynPort Vaccine Company, a CSC Company
Locations (11):
- United States (11):
  - Benchmark Research, San Francisco, California
  - Apex Research Institute, Santa Ana, California
  - Johnson County Clinical Trials, Lenexa, Kansas
  - Heartland Reseach Assoicates, LLC, Wichita, Kansas
  - Central Kentucky Research Associates, Lexington, Kentucky
  - WRAIR Clinical Trials Center, Silver Spring, Maryland
  - Center for Pharmceutical Research, Kansas City, Missouri
  - Rochester Clinical Research, Rochester, New York
  - Wake Research Associates, Raleigh, North Carolina
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - New Orleans Center for Clinical Research, Knoxville, Tennessee